CLINICAL TRIAL: NCT06248008
Title: An Open, Multicenter, Phase III Extension Clinical Trial to Evaluate the Long-term Safety of ASC40 (Denifanstat) Tablets in Patients With Moderate to Severe Acne Vulgaris
Brief Title: A Study to Evaluate Safety of ASC40 Tablets in Patients With Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC40-304
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Acne
Keywords: Acne; ASC40
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASC40 50mg (Experimental): ASC40 50mg, up to 40 weeks of treatment.
  Interventions: Drug: ASC40

INTERVENTIONS:
Drug: ASC40 — ASC40 tablets orally once daily

SUMMARY:
This is a multicenter, open-label study designed to determine the long-term safety of ASC40 (Denifanstat) tablets in patients with moderate to severe acne vulgaris enrolled in the ASC40-303 Phase III study. All subjects are eligible for study eligibility screening after enrollment in ASC40-303 Phase III study, and all eligible subjects with moderate to severe acne vulgaris will receive ASC40 (Denifanstat) tablets after signing informed consent. The investigational drug will be administered orally once daily (QD) for up to 40 weeks. There will be a total of 7 visits for screening and follow-up. The tests required by the program included routine blood tests, blood biochemistry, lipid profile, pregnancy test and urine routine, etc.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have successfully completed a 12-week Phase III study of ASC40-303;
* Have fully understood this research and voluntarily signed the informed consent;
* The fertile male and female subjects of reproductive age agreed to use effective contraception from the time they signed the informed consent until 3 months after the final administration of the investigationa drug;
* Subjects are willing and able to complete the study, understand and comply with the study requirements, comply with the study requirements restrictions and related education, use the investigational drug as prescribed by the physician, and follow up according to the study schedule.

Exclusion Criteria:

* Discontinue participation in the ASC40-303 Phase III study for any reason;
* Are receiving/planning to receive any systemic acne medications, systemic retinoids, systemic corticosteroids, or any androgen/antiandrogen therapy (e.g., testosterone, spironolactone);
* Pregnant, nursing, or planning a pregnancy during the study period;
* Have major complications (including clinically significant abnormalities in clinical laboratory tests), mental disorders, or other factors deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects with treatment emergent adverse events (TEAE) | From the first dose to 40 weeks of treatment.
  The number and percentage of all subjects with treatment emergent adverse events (TEAE) from the first dose to 40 weeks of treatment.
Number and percentage of subjects with serious adverse event (SAE). | From the first dose to 40 weeks of treatment.
  Number and percentage of subjects with serious adverse event (SAE) from the first dose to 40 weeks of treatment.
Number and percentage of subjects who discontinued due to adverse events. | From the first dose to 40 weeks of treatment.
  Number and percentage of subjects who discontinued due to adverse events from the first dose to 40 weeks of treatment.

SECONDARY OUTCOMES:
At the end of the visit, the number of people whose IGA rating had decreased by at least 2 points from the baseline period of the study. | up to 40 weeks.
  At the end of the visit, the number of subjects whose IGA rating had decreased by at least 2 points from the baseline period of the study.
At the end of the visit, the number of subjects with an IGA score of 3 or higher at baseline dropped to an IGA score of 0 or 1. | up to 40 weeks.
  At the end of the visit, the number of subjects with an IGA score of 3 or higher at baseline dropped to an IGA score of 0 or 1 among all subjects.
Percentage change in total skin lesion count at the end of the visit compared to the baseline period of the study. | up to 40 weeks.
  Percentage change in total skin lesion count at the end of the visit compared to the baseline period of the study.
Percentage change in total inflammatory skin lesion count at the end of the visit compared to the baseline period of the study. | up to 40 weeks.
  Percentage change in total inflammatory skin lesion count for all subjects at the end of the visit compared to the baseline period of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China